CLINICAL TRIAL: NCT05819788
Title: Outcomes of Fresh Frozen Plasma Usage During Cardiopulmonary Bypass in Congenital Cardiac Surgery.
Brief Title: FFP Usage in Pediatric CV Surgery
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00129275
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Coagulopathy; Congenital Heart Disease
MeSH Terms: conditions — Hemostatic Disorders; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FFP: Patients undergoing CPB receiving FFP
- no FFP: Patients undergoing CPB not receiving FFP

SUMMARY:
When small children undergo heart surgery with the heart-lung machine, in the past, blood products to help the blood clot such as Fresh Frozen Plasma (FFP) was routinely used in children under 10kg. With blood clot monitoring technology, we feel that it might not be necessary to expose all children to FFP. We want to determine if those children who did not receive FFP bleed more or require more blood products as compared to those who did receive FFP while on the heart lung machine.

DETAILED DESCRIPTION:
This will be a single center, retrospective study. Our cohort will include pediatric patients between 4 and 8 kilograms undergoing congenital cardiac surgery with cardiopulmonary bypass between January 2019 and January 2023. Patients will be divided into two groups: FFP given at onset of CPB and no FFP given intraoperatively. Patients requiring FFP for heparin resistance and anti-thrombin III deficiency will be excluded. Patient clinical, surgical, and bypass characteristics, transfusion, and bleeding outcomes will be collected using REDCAP and via chart review using Connect Care.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients between 4 and 8 kilograms undergoing congenital cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Patients requiring FFP for heparin resistance and anti-thrombin III deficiency will be excluded

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: pediatric patients between 4 and 8 kilograms with congenital cardiac defects
Sampling Method: Non-Probability Sample
Enrollment: 431 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Transfusion | 24 hours
  Units of blood products transfused
Bleeding | 24 hours
  Chest tube output

SECONDARY OUTCOMES:
Length of ventilation | 5 days
  Time to extubation
Length of stay | 5 days
  Time to ICU ready for discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mancho Ng, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada